CLINICAL TRIAL: NCT01195480
Title: Immunotherapy With CD19ζ Gene-modified EBV-specific CTLs After Stem Cell Transplant in Children With High-risk Acute Lymphoblastic Leukaemia
Brief Title: CD19-CAR Immunotherapy for Childhood Acute Lymphoblastic Leukemia (ALL)
Acronym: CD19TPALL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to lack of biological efficacy and CD19 CAR CTL persistence
Sponsor: University College, London (Other)
Collaborators: European Union (Other); The Leukemia and Lymphoma Society (Other); Children with Leukaemia (Unknown); Department of Health, United Kingdom (Other Government); JP Moulton Charitable Foundation (Other); Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/09/0050; 2007-007612-29 (EudraCT Number)
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Immunotherapy; Gene Therapy; Paediatric; B cell Acute Lymphoblastic Leukaemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylaxis arm (Experimental): Patients who have relapsed in the bone marrow after previous myeloablative HSCT and achieve remission after chemotherapy will be treated prophylactically with CD19-specific gene-engineered T cells after a second HSCT with reduced intensity conditioning.
  Interventions: Genetic: donor-derived EBV-specific cytotoxic T-cells (EBV-CTL) transduced with the retroviral vector SFGalpha-CD19-CD3zeta; Biological: Irradiated donor-derived Lymphoblastoid Cell Line
- Pre-emptive arm (Experimental): In this arm, patients identified at high (> 50%) risk of relapse will be eligible for generation of donor-derived EBV CTL immediately prior to HSCT. These patients will be monitored for evidence of MRD in regular bone marrow aspirates for the first year post-HSCT. MRD positivity post-HSCT is highly predictive of subsequent relapse. In those patients who become MRD+ in the marrow at a level of minimum 5 x 10-4, cryopreserved CTL that have been transduced with a retroviral vector carrying the CD19-zeta transgene will be thawed and administered to the patient pre-emptively.
  Interventions: Genetic: donor-derived EBV-specific cytotoxic T-cells (EBV-CTL) transduced with the retroviral vector SFGalpha-CD19-CD3zeta; Biological: Irradiated donor-derived Lymphoblastoid Cell Line

INTERVENTIONS:
Genetic: donor-derived EBV-specific cytotoxic T-cells (EBV-CTL) transduced with the retroviral vector SFGalpha-CD19-CD3zeta — All patients will be treated at the same total dose level of 2 x 10^8/m2
Biological: Irradiated donor-derived Lymphoblastoid Cell Line — The initial cohort of 5 patients (regardless of arm of study) will be treated as described. If transduced CTL infusion is safe in this initial cohort and real-time DNA PCR studies demonstrate that transduced CTL are undetectable in > 50% of patients by 2 months post-infusion, the remaining 25 patients (in either arm of the study) will be treated as above but with an additional vaccination of CD19-zeta-transduced EBV-LCL infusion.
  Vaccination will consist of 3 doses of 5 x 10^6 irradiated (70Gy) donor-derived EBV-lymphoblastoid cell line used to generate CTL and will be administered subcutaneously into the thigh (volume 0.3 ml) at day -2, week 4 and 8 post-transduced CTL infusion.

SUMMARY:
The aim of this clinical trial is to evaluate the feasibility, safety and biological effect of adoptive transfer of CD19ζ chimaeric receptor transduced donor-derived EBV-specific cytotoxic T-lymphocytes (EBV-CTL) in patients with high-risk or relapsed B cell precursor ALL after allogeneic Haematopoietic Stem Cell Transplantation (HSCT).

ELIGIBILITY:
Inclusion Criteria Pre-emptive arm

Children (18 years or younger) with CD19+ precursor B cell ALL fulfilling one of the following criteria who are undergoing an allogeneic stem cell transplant from an EBV-seropositive donor:

In first remission, if at least one of the following criteria are met:

* t(9;22) and MRD positive (BCR-ABL/ABL ratio > 0.01%) after HR3 block of EsPhALL or pre-HSCT or
* Infant ALL age < 6 months at diagnosis with MLL gene rearrangement and either presenting wcc >300 x 10^9/L or poor steroid early response (i.e circulating blast count >1x10^9/L following 7 day steroid pre-phase of Interfant 06) or
* Resistant disease (> 30% blasts at end of induction treatment day 28-33) in subsequent morphological CR or
* High level bone marrow MRD (> 1 in 1000) at week 12 ALL-BFM 2000/AIEOP BFM ALL 2009/EORTC 58951 protocols, week 12-15 of FRALLE A or at week 14 of UKALL2011

Relapsed patients if at least one of the following criteria are met:

* Very early (< 18 months from diagnosis) bone marrow or extramedullary relapse in second CR or
* Early (within 6 months of finishing therapy) isolated bone marrow relapse with bone marrow MRD > 1 in 100 at day 35 of reinduction in second CR or
* Early (within 6 months of finishing therapy) bone marrow or combined relapse with high level bone marrow MRD (> 1 in 1000) at the end of consolidation therapy (week 12-13 UKALL R3/INTREALL and COOPRALL protocols, prior to protocol M in BFM relapse protocol (ALL-REZ BFM 2002) and after Protocol II-IDA in AIEOP LLA Rec 2003)or
* Any relapse of infant or Philadelphia-positive ALL in morphological complete remission
* Any patient being transplanted in 3rd or greater CR

These patients have a high (> 50%) risk of relapse and will be monitored for evidence of MRD in bone marrow aspirates (monthly for months 1-6, 6 weekly months 7.5-12 post HSCT) for the first year post-transplant. Patients who become MRD +ve in the marrow at a level minimum 5 x 10-4 (or BCR-ABL/ABL ratio 0.05% in Ph+ve ALL patients with no IgH MRD marker) but are in morphological remission (<5% blasts in BM) will be eligible to be treated pre-emptively with CD19ζ transduced CTL

Prophylaxis arm

Additionally, any patient (≤ 18 years) with ALL relapsing in the bone marrow (isolated or combined) after myeloablative allogeneic HSCT who achieves morphological remission after re-induction and who is a candidate for second HSCT at one of the participating centres is eligible to receive CD19ζ transduced CTL prophylactically

* Stem cell donors must be EBV sero-positive and HLA-matched (8/8 HLA A,B,C and DR at medium resolution typing) or a single antigenic/allelic (7/8) mismatch with the recipient
* A life expectancy of at least 12 weeks
* Karnofsky score of >60% if >10 years old or Lansky performance score of >60 if ≤ 10 years old
* Patients must have transduced donor-derived EBV-specific CTLs with 15% or higher expression of CD19ζ determined by flow-cytometry which meet the specified release criteria
* Informed written consent indicating that patients are aware this is a research study and have been told of its possible benefits and toxic side effects

Exclusion Criteria

* Patients with CD19 negative precursor B cell ALL
* EBV seronegative or > single antigenic/allelic HLA-mismatched donor
* Active acute GVHD overall Grade 2 or higher or significant chronic GVHD requiring systemic steroids at the time of scheduled infusion of transduced CTL will be excluded until the patient is GVHD-free and off steroids
* Pre-existing severe lung disease (FEV1 or FVC < 50% predicted) pre-HSCT or an oxygen requirement of >28% O2 supplementation or active pulmonary infiltrates on chest X-ray at the time scheduled for transduced CTL infusion
* Serum bilirubin >3 times the upper limit of normal or an AST or ALT > 5 times the upper limit of normal
* Serum creatinine >3 times upper limit of normal
* Active severe intercurrent infection at the time of transduced CTL infusion (if present consult with Chief investigator).
* Patients in whom transduced donor-derived EBV-specific CTLs don't meet release criteria
* Serologically positive for Hepatitis B, C or HIV pre-HSCT
* Females of childbearing age with a positive pregnancy test
* Known allergy to DMSO

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2012-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Toxicity attributable to transfer of CD19-zeta transduced CTL | 1 year
  1. Incidence of grade 3-5 toxicity attributable to transfer of CD19-zeta transduced CTL within 12 weeks of infusion.
  2. Incidence of significant (Grade II-IV) and severe (Grade III-IV) acute GVHD before day 100 and limited/extensive chronic GVHD between day 100-365.
  3. Incidence of hypogammaglobulinaemia after CD19-zeta CTL transfer at day 100, 6 months and 1 year post-HSCT
Biological efficacy as assessed by effect of CD19-zeta transduced CTL on Minimal Residual Disease levels in the bone marrow in the first year post- transduced CTL infusion | 1 year

SECONDARY OUTCOMES:
Persistence and frequency of circulating CD19-zeta transduced CTL in the peripheral blood of recipients after adoptive transfer as assessed by flow cytometry and quantitative real-time PCR. | 1 year
In vitro anti-leukaemic response of circulating PBMC post adoptive transfer of CD19-zeta transduced CTL using interferon-gamma ELISPOT assays after stimulation with CD19+ve targets | 1 year
Relapse rate, disease-free survival and overall survival at 1 and 2 years after adoptive immunotherapy with CD19ζ-transduced EBV-CTL | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Persis Amrolia, Professor, Study Chair — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (7):
- Germany (4):
  - Klinik und Poliklinik für Kinder- und Jugendmedizin, Universitätsklinikum, Essen
  - Hospital for Children and Adolescents III, Goethe University, Frankfurt
  - Medizinische Hochschule, Hanover
  - University Children's Hospital, Münster
- United Kingdom (3):
  - Bristol Children's Hospital, Bristol
  - Great Ormond Street Hospital for Children, London
  - University College London Hospital, London

REFERENCES:
- See also: Final Publication — http://www.nature.com/leu/journal/vaop/ncurrent/full/leu201739a.html